CLINICAL TRIAL: NCT01951989
Title: Study of Intra-monocytic Imiglucerase Kinetic and Its Correlation With Clinical and Biological Gaucher Disease
Brief Title: Intra-monocyte Imiglucerase Kinetics in Gaucher Disease
Acronym: CIMI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0167; 2012-019622-13
Record Dates: First submitted 2013-09-02; First posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease; Imiglucerase; Pharmacokinetics
MeSH Terms: conditions — Gaucher Disease | interventions — Pharmaceutical Preparations; Pharmacokinetics

ARMS (1):
- Imiglucerase (Experimental): Primary purpose: to evaluate the pharmacokinetics of Imiglucerase activity into target cellular compartment depending on dose and frequency of infusions.
  Secondary purposes : 1) to establish a possible relationship between the intra-monocytic activity of glucocerebrosidase and the clinical and biological activity of Gaucher disease and to define a possible threshold value of enzyme activity; 2) to establish a better correlation with known biomarkers of disease (routine markers and markers recently identified), which would better predict and / or monitor response to treatment ; 3) to compare the residual and natural rate of activity enzyme intra-monocytic for untreated patients (low severity disease).
  Interventions: Drug: Imiglucérase (drug) pharmacokinetics

INTERVENTIONS:
Drug: Imiglucérase (drug) pharmacokinetics

SUMMARY:
Rational: Imiglucerase has been used to treat Gaucher disease since 1997 but data about its pharmacokinetics have been partial; investigators know that imiglucerase undergoes a quick clearance from plasma compartment following the infusion (1/2 life: 1-6 min, from tissue: <24h), an observation apparently contradictory with usual infusion rhythm (one infusion every two weeks). Furthermore, by going by GD response, the rhythm of Infusion is sometimes diminished (for example, every 3 or 4 wks) without pharmacological rational ; In parallel, investigators demonstrated that monocytes represent a satisfactory surrogate of GD target cells and that enzyme activity into monocytes varies between individuals.

Our hypothesis is that enzyme activity into monocyte compartment could be different and could be related to GD response.

Primary purpose: to evaluate the pharmacokinetics of Imiglucerase activity into target cellular compartment depending on dose and frequency of infusions.

Secondary purposes : 1) to establish a possible relationship between the intra-monocytic activity of glucocerebrosidase and the clinical and biological activity of Gaucher disease and to define a possible threshold value of enzyme activity; 2) to establish a better correlation with known biomarkers of disease (routine markers and markers recently identified), which would better predict and / or monitor response to treatment ; 3) to compare the residual and natural rate of activity enzyme intra-monocytic for untreated patients (low severity disease).

DETAILED DESCRIPTION:
Rational: Imiglucerase has been used to treat Gaucher disease since 1997 but data about its pharmacokinetics have been partial; investigators know that imiglucerase undergoes a quick clearance from plasma compartment following the infusion (1/2 life: 1-6 min, from tissue: <24h), an observation apparently contradictory with usual infusion rhythm (one infusion every two weeks). Furthermore, by going by GD response, the rhythm of Infusion is sometimes diminished (for example, every 3 or 4 wks) without pharmacological rational ; In parallel, investigators demonstrated that monocytes represent a satisfactory surrogate of GD target cells and that enzyme activity into monocytes varies between individuals. Our hypothesis is that enzyme activity into monocyte compartment could be different and could be related to GD response.

Primary purpose: to evaluate the pharmacokinetics of Imiglucerase activity into target cellular compartment depending on dose and frequency of infusions.

Secondary purposes : 1) to establish a possible relationship between the intra-monocytic activity of glucocerebrosidase and the clinical and biological activity of Gaucher disease and to define a possible threshold value of enzyme activity; 2) to establish a better correlation with known biomarkers of disease (routine markers and markers recently identified), which would better predict and / or monitor response to treatment ; 3) to compare the residual and natural rate of activity enzyme intra-monocytic for untreated patients (low severity disease).

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 12 years old with Gaucher disease type 1 or type 3 and having signed an informed consent
* Treated with imiglucerase (Cerezyme ®) with a stable therapeutic strategy for at least 3 months.

OR

* Untreated patient, with no therapeutic indication at the time of inclusion and having a diagnosis older than 2 years (non progressive disease)
* Patients must have a social security system

Exclusion Criteria:

* Age <12 years old
* Gaucher disease unproven
* Gaucher disease treated with therapeutic changes in the previous 3 months, or current treatment different from imiglucerase
* Gaucher disease untreated whose diagnosis was established for under 2 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-02 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Enzyme intra-monocyte activity (sum of endogenous enzyme activities and therapeutic enzyme)in patients treated with imiglucerase | at day 1
  Enzyme intra-monocyte activity (sum of endogenous enzyme activities and therapeutic enzyme) in patients treated with imiglucerase will be assessed at different times between infusions (8 to 10 time points), and just before an infusion (residual rate). The population pharmacokinetics method allows to perform this analysis in measurement windows that are not necessarily included in the period between two consecutive infusions of imiglucerase but may be spread over several cycles.

SECONDARY OUTCOMES:
Residual rate | every 6 months during 2 years.
  Pharmacokinetics descriptive criteria are the area under curve at balance, the terminal half-life and the residual rate.
Endogeneous intra-monocyte glucocérébrosidase activity from untreated patients | every 6 months during 2 years
Biomarker dosages will provide serum concentration values | at D0, M3, M6 and every 6 months during 2 years:
  1) routine biomarkers (ACE, TRAP, chitotriosidase, ferritin) and 2) potentially interesting biomarkers but not routinely evaluated in France (CCL18, MIP1a, MIP1b, MCP1, IL-8, glycated ferritin).
  - Gaucher disease status will be assessed by clinical and biological criteria defined by the HAS (Haute Autorité de Santé = High Health Authority). We will consider the two-year periods before and after treatment to identify progressive diseases (clinical or biological significant events associated with Gaucher disease in the two years before and 2 years after the enrolment time

CONTACTS AND LOCATIONS:
Overall Officials: Marc BERGER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France